CLINICAL TRIAL: NCT01859507
Title: Study of the Effectiveness and Safety of Clostridium Botulinum Type A Neurotoxin Complex Injection in the Perineal Muscles in Resistant Cases of Vaginismus
Brief Title: Injection of Botox in the Perineal Muscles in Resistant Cases of Vaginal Spasm
Acronym: VginsmsBOTOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdel-Maguid Ramzy (Other)
Responsible Party: Sponsor-Investigator, Abdel-Maguid Ramzy, Prof. Of OB. GYN.,, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ramzy9501
Record Dates: First submitted 2013-05-19; First posted 2013-05-22 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Vaginismus
Keywords: Vaginismus; Botox; Sex; Clostridium; Botulinum; Neurotoxin; Perineal; Muscles
MeSH Terms: conditions — Vaginismus; Coitus | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BOTOX group (Experimental): Injection of BOTOX in the perineal muscles in resistant cases of vaginismus. Proper informed consent forms will be signed. The injection procedure is done under local anesthesia for most of our patients. We followed up the patient by phone calls for possible adverse effects following the procedure for 4 days.The patient is then instructed to attend dilatation sessions twice weekly in the clinic, in the presence of the husband, for 3-4 weeks. We use silicone dilators, of ascending sizes, covered by lubricated condoms. In the initial phase of the dilatation procedure we start each session with the appropriate size of the dilator according to the capacity of the introitus and the degree of vaginismus, and thereafter increase the size gradually.
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — In the first session, proper history taking and proper counseling of the couple including the description of the new modality (BOTOX injection) of treatment and subsequent dilatation sessions. During examination, all our maneuvers are gentle to gain trust of the patient. Following sterilization, we used surface (Xylocaine gel 2% ASTRA ZENECA) anesthesia before the injection. In addition we used finger like ice packs pre-prepared in a surgical latex glove, on the perineum. We made sure to check that the tip of the needle is not in a vessel by aspirating before proceeding with the injection of each bolus of BOTOX.
  Other Names: Clostridium Botulinum type A neurotoxin complex

SUMMARY:
During the first visit, the couple will be acquainted with their condition. This will include the epidemiology of their condition, some sex education tips, as well as the therapeutic modalities available. This is followed by short description of the protocol. In the procedure room, each patient will be examined to determine the degree of vaginismus and classify her condition according to Lemont's classification as modified by Pacik, from 1 to 5. In the same or subsequent sessions, surface anesthesia of the area of injection followed by ice packs is used before the BOTOX is injected into the muscle.

DETAILED DESCRIPTION:
In the first session, proper history taking includes the difficulties they are facing, and the measures taken to solve it whether medical or folk treatment. Proper counseling of the couple to describe the new modality including the BOTOX injection and subsequent dilatation sessions. Proper informed consent forms will be signed. Therapy sessions will starts with the gentle informed approach to the genital area to gain trust of the patient. This is followed by the digital vaginal examination of the patient to determine the degree of spasm and the muscle(s) involved.

The patient will be asked to lie down comfortably on the examination table in the lithotomy position. Her husband is allowed to stand on her left shoulder side and may be allowed to hold her hand. We started by sterilizing the perineal area and injection site in the vaginal introitus using povidone iodine solution. The patient is warned effectively before each step of the procedure and what to expect as regards pain. We used surface (Xylocaine gel) anesthesia half an hour before the injection.We did not use local anesthetic infiltration injections at the site of BOTOX injection. In addition we used ice packs, pre-prepared in a surgical latex glove finger, on the perineum and introitus before the injection of BOTOX to act as a counter irritant. However in advanced cases of Vaginismus (V4-5), we used general intravenous anesthesia

We made sure to check that the tip of the needle is not in a vessel by aspirating before proceeding with the injection of each bolus of BOTOX. We only did one skin puncture, and used that to radially injecting the intended area by changing the direction of the tip of the needle. We found this much less painful to the patient. The injection site will be monitored by the other free hand index and thumb. Following the withdrawal of the needle from the muscle, we distributed the bolus of BOTOX uniformly within the muscle digitally using an arc fashion massage of the introitus. We applied pressure, whenever needed to stop the bleeding from the injection site.

Following the procedure, we instruct the patient to do Kegel exercises as much as 100 contractions or more over 48 hours. This will help in distributing the BOTOX within the muscles as well as recognition of the patient of the whereabouts of the muscles involved in vaginismus. We followed up on our patients daily by phone calls for 4 days following the procedure for possible adverse effects.

Thereafter, the patient will be instructed to attend dilatation sessions twice weekly in the clinic, in the presence of the husband, for 3-4 weeks. We use silicone dilators covered by lubricated condoms. We prepared the vaginal introitus by the use K-Y jelly for lubrication of the dilators. The patient is introduced to the dilator and allowed to hold it in her hand, for size and feel, prior to its introduction into her vagina. During each session the patient will be asked to lie down on the examination table in the lithotomy position, relax and feel comfortable. The husband may stand beside her and may hold her hand. In the initial phase of the dilatation procedure we start with the appropriate size of the dilator according to the capacity of the introitus and the degree of vaginismus, in each session, and increase the size gradually. We always start by the smaller size and move up size wise. At later sessions we allow the patient herself with its introduction into the vagina using only her tactile sense, with no visual aid or doctor instructions, covering her thighs with sheets to feel more private. She is asked to report the termination of the introduction or difficulties she is facing. Verbal support is always and repeatedly used. In case of difficulty, the doctor does not offer to help and ask the patient to try on her own once more. This helps her to be proactive and gain control of the procedure. They usually succeed to carry on the procedure on their own. The couple will be instructed not to have trials of intercourse before the patient uses dilator number 4 comfortably.

ELIGIBILITY:
Inclusion Criteria:

* cases with resistant vaginismus

Exclusion Criteria:

* cases with congenital anomalies in the lower female genital tract

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbdelMaguid I Ramzy, MD, Principal Investigator — Cairo University
Locations (1):
- AbdelMaguid Ramzy, Cairo, Egypt

REFERENCES:
- [Background] Pacik PT. Vaginismus: review of current concepts and treatment using botox injections, bupivacaine injections, and progressive dilation with the patient under anesthesia. Aesthetic Plast Surg. 2011 Dec;35(6):1160-4. doi: 10.1007/s00266-011-9737-5. Epub 2011 May 10. PMID 21556985
- See also: Botox Injection for Treatment of Vaginismus. Peter T. Pacik — http://clinicaltrials.gov/ct2/show/NCT01352546

RESULTS

PARTICIPANT FLOW:
Groups:
- Botox: Injection of Clostridium Botulinum type A neurotoxin complex in the perineal muscles in resistant cases of vaginismus.
  Trade Name:
  BOTOX 100 units vial
  Injection of Botox in the perineal muscles in resistant cases of vaginismus
Period: Overall Study
Arm/Group | Botox
Started | 32
Completed | 28
Not Completed | 4
Not completed — left the country | 4

BASELINE CHARACTERISTICS:
Population: All participants who completed the study
Arm/Group | Botox
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.25 (4.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 28

OUTCOME MEASURES:

1. Primary Outcome: Success of Repeated Penetration of the Penis Through the Vaginal Introitus Into the Vagina Without or With Acceptable Pain
Description: The primary outcome will be assessed by the couple. The couple is allowed to visit for follow up in a 4 weeks' time. Our inquiry is on the success of full and repeated penetration of the penis through the vaginal introitus into the vagina without or with acceptable pain. An acceptable outcome will be at least twice weekly successful sexual relationship that was completed without premature interruption from either partners.
Time Frame: Up to four weeks following the last session of the vaginal dilatation.
Population: multiple penetration with minimal pain as informed by the couple during their follow up sessions 4 weeks after the completion of the dilatation sessions
Measure: Number; unit: participants
Arm/Group | Botox
Number analyzed (Participants) | 28
participants | 28

2. Secondary Outcome: Successful Sexual Relationship
Description: The level of comfort by the couple. The secondary outcome will be assessed by the couple. The couple is allowed to visit for follow up every three months for twelve months. Our inquiry is on the success of full and repeated penetration of the penis through the vaginal introitus into the vagina without or with acceptable pain. An acceptable outcome will be at least twice weekly successful sexual relationship that was completedwithout premature interruption from either partners.
Time Frame: Within twelve months after the Botox injection
Measure: Number; unit: participants
Groups:
- BOTOX Group: Injection of BOTOX 100 units vial as a single dose intramuscular in the perineal muscles. Proper informed consent forms will be signed. In most of the cases we use local anesthetic before injection. However in V4 and 5 we resort to general anesthesia. We followed up the patient by phone calls daily for possible adverse effects following the procedure for 4 days, which is the interval allowed for the BOTOX to be fully effective. The patient is then instructed to attend dilatation sessions twice weekly in the clinic, in the presence of the husband, for 3-4 weeks. We use silicone dilators covered by lubricated condoms. We start each session with the appropriate size of the dilator according to the capacity of the introitus and increase the size gradually thereafter. We proceed till the patient uses the largest dilator with no or limited pain. The patient is then advised then to try to have intercourse and report back to us.
  Botox: In the first session, proper histor
Arm/Group | BOTOX Group
Number analyzed (Participants) | 28
participants | 28

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: 2 participants who started the study could not be reached for adverse event monitoring. Participants were monitored for 4 days closely for adverse events related to the injection and then via phone for a year for any additional adverse events.
Arm/Group | Botox
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes